CLINICAL TRIAL: NCT04066738
Title: SCar Location and Acute Haemodynamic Response to MultiPoint Pacing in Patients With Ischemic Cardiomyopathy (SCAR MPP Study)
Brief Title: Scar Location and Acute Haemodynamic Response to MultiPoint Pacing Study in Patients With Ischemic Cardiomyopathy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to recruit
Sponsor: Oxford University Hospitals NHS Trust (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Principal Investigator, Tim Betts MD MBChB FRCP, Principle Investigator, Consultant Cardiologist, Oxford University Hospitals NHS Trust
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12193
Record Dates: First submitted 2019-04-17; First posted 2019-08-26 (Actual); Results first posted 2022-05-18 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-03

CONDITIONS: Heart Failure; Ischemic Cardiomyopathy
Keywords: MultiPoint Pacing; Acute Haemodynamic Response
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with myocardial scar (Other): Patient with previous STEMI resulting in myocardial scar, elected to CRT implant
  Interventions: Diagnostic Test: Cardiac MRI with gadolinium contrast; Diagnostic Test: 3D reconstruction and location of coronary sinus venous system relative to myocardial scar; Diagnostic Test: Acute haemodynamic measurements during CRT implant

INTERVENTIONS:
Diagnostic Test: Cardiac MRI with gadolinium contrast — Imaging of left ventricular scar and coronary sinus venous system
Diagnostic Test: 3D reconstruction and location of coronary sinus venous system relative to myocardial scar — Three dimensional mapping of coronary sinus venous system with Abbott Precision mapping system and Biotronik Vision wire Merge with MRI images of CS and myocardial scar
Diagnostic Test: Acute haemodynamic measurements during CRT implant — Advancement of pressure wire to LV cavity via femoral/radial arterial access. Real time measurement of LV-dP/dTmax during conventional CRT and MPP after consecutive placement of LV lead in two different CS branches (peri-infarct region and remote myocardium)

SUMMARY:
Cardiac Resynchronization Therapy (CRT) is a proven treatment for heart failure.

CRT consists of a special pacemaker with two/three leads (insulated wires which take the electrical impulses from the device to the heart), one in the right ventricle, one in a vein on the outer surface of the left ventricle (in a vessel called coronary sinus or CS) and sometimes one in the right atrium (right top chamber of the heart). Tiny electrical impulses are simultaneously sent to the ventricles to make them beating together again in a more synchronised pattern. This leads to a coordinated, synchronous pumping action that, in most patients, translates into improved heart failure symptoms and improved quality and quantity of life, reducing the chance of being admitted to hospital with worsening heart failure. Unfortunately up to one third of the patients do not benefit from CRT therapy and to date there are no useful criteria to predict the response to CRT.

In an effort to improve the response rate to CRT, alternative methods have been developed. In particular, a new technology called MultiPoint Pacing (MPP) (St. Jude Medical, Sylmar, CA) has recently become available. It allows simultaneous stimulation of 2 different points in the left ventricle by using a single lead with four electrodes. This strategy should improve the pumping function of the heart by recruiting a larger mass of muscle. Although MPP is as safe and as effective as standard CRT pacing, the improvements to date in the heart pump function it gives over standard CRT pacing are variable and small.

Recent evidence suggests that MPP pacing could be particularly beneficial in some subgroups of patients, in particular patients with a previous history of heart attack resulting in scar formation in the left ventricle.

The investigators hypothesize that MPP works better when the lead is closer to the scar because this allows recruitment of areas with slow conduction, thus increasing synchronization further.

To this aim, they plan to compare, in each patient, the acute response produced by MPP on the cardiac function when the CS lead is placed close to myocardial scar and when it is placed far from scar respectively.

DETAILED DESCRIPTION:
A prospective single-centre pilot study will be conducted to investigate this topic. Fifteen patients, with a history of previous ST Elevation Myocardial Infarction (STEMI) resulting in myocardial scar and elected to CRT implant at the OUH, will be enrolled in this study.

Compared to standard practice, additional research investigations will be a baseline visit for eligibility assessment, informed consent and pre-CRT implant cardiac MRI, a three-dimensional electroanatomical map reconstruction of the CS venous system during the standard CRT implant and the evaluation of the acute haemodynamic response (AHR, percentage increase of LV-dP/dT max) of MPP over conventional single-site LV pacing during the CRT implant.

The cardiac Magnetic Resonance Imaging (MRI) will be performed in each patient 1-2 weeks before the CRT implant during the baseline visit. It will provide information regarding presence and location of myocardial scar and anatomy of the CS venous system.

A de-novo CRT implant will be performed under fluoroscopic guidance as per standard care. All subjects will be implanted with a regulatory approved St. Jude Medical CRT device compatible with MPP feature (models n° CD3271-40(Q), CD3371-40(Q), CD3371-40C(QC) or newer) and St. Jude Medical quadripolar left ventricular lead (Quartet 1458Q or newer). The choice of the right ventricular and right atrial leads will be left to the operator. After implant of the right ventricular and right atrial leads, a CS venogram will be then performed as per standard practice (see intervention section for more details).

A three-dimensional electroanatomical map of the CS venous system will be constructed with Precision mapping system and a Biotronik Vision wire (Biotronik Se & Co. KG, Berlin, Germany) by using the CS venogram as a guide. The map will be merged with the correspondent cardiac MRI images in order to locate the myocardial scar in respect to the CS branches. This will allow the identification of two target CS branches for the study measurements, one located in the peri-infarct region and one located in the remote myocardium.

A Certus PressureWire will be then introduced into the LV. A PhysioMon software (Radi Medical Systems, Uppsala, Sweden) will be used for electronic calculation of the LV-dP/dTmax from every heartbeat for a period of at least thirty seconds to ensure steady-state conditions. The baseline LV-dP/dTmax will be measured during ventricular spontaneous rhythm.

A St. Jude Medical quadripolar left ventricular lead will be sequentially placed in the "peri-infarct" CS branch and in the "remote myocardium" CS branch. In each site the percentage increase in LV-dP/dTmax (Acute Haemodynamic Response, AHR) produced by both conventional single-site and MPP LV pacing to will be measured. All 4 poles of the quadripolar lead will be used in turn for conventional single-site LV pacing, 3 different configurations will be used in turn for MPP. The LV-dP/dTmax will be recorded for each pacing configuration in order to identify the MPP and the single-site LV pacing configurations producing the best AHR (best percentage increase of LV-dP/dTmax).

The AHR produced by the best MPP configuration in peri-infarct region will be compared with the AHR produced by the best MPP configuration in the remote myocardium. Moreover, the percentage increase of LV-dP/dTmax produced by the best MPP configuration over the best conventional single-site LV pacing in the peri-infarct region will be compared with the same measurement obtained in the remote myocardium.

The decision about the final position of the LV lead and the activation of MPP feature after the CRT implant will be left to operator preference.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 years or over
* Previous STEMI (> 3 months before enrolment) and consequent LV scar;
* Standard indication to CRT-D (NYHA functional class III-IV despite optimal medical therapy, LV ejection fraction (LVEF) ≤35 %, QRS duration ≥120 msec, LBBB);
* Sinus rhythm;
* Will and ability to give informed consent for participation in the study.

Exclusion Criteria:

* Pregnancy, trying for a baby or breast feeding;
* Any other significant disease or disorder which, in the opinion of the investigator, may either put the participants at risk because of participation in the study, or may influence the result of the study, or the participant's ability to participate in the study;
* Inability to tolerate MRI scanning (e.g. claustrophobia, unable to lie flat)
* Contraindications to MRI scanning (e.g. implantable devices, cranial aneurysm clips, metallic ocular foreign bodies, hypersensitivity to gadolinium);
* Significantly impaired renal function (eGFR < 30ml/min);
* History of allergy to cardiac MRI contrast media;
* Severe claustrophobia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2017-09-27 (Actual); Primary Completion 2017-10-23 (Actual); Study Completion 2020-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tim Betts, MD, Principal Investigator — Oxford University Hospitals NHS Trust
Locations (1):
- John Radcliffe Hospital, Oxford, United Kingdom

RESULTS

PARTICIPANT FLOW:
Groups:
- Patients With Myocardial Scar: Patient with previous STEMI resulting in myocardial scar, elected to CRT implant
  Cardiac MRI with gadolinium contrast: Imaging of left ventricular scar and coronary sinus venous system
  3D reconstruction and location of coronary sinus venous system relative to myocardial scar: Three dimensional mapping of coronary sinus venous system with Abbott Precision mapping system and Biotronik Vision wire Merge with MRI images of CS and myocardial scar
  Acute haemodynamic measurements during CRT implant: Advancement of pressure wire to LV cavity via femoral/radial arterial access.
  Real time measurement of LV-dP/dTmax during conventional CRT and MPP after consecutive placement of LV lead in two different CS branches (peri-infarct region and remote myocardium)
Period: Overall Study
Arm/Group | Patients With Myocardial Scar
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Patients With Myocardial Scar
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 2
Age, Continuous [Mean (Standard Deviation); unit: years] — Age at the time of enrolment, measured in years
  years | 65 (2.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United Kingdom | 2
dP/dt produced by MPP in the peri-infarct region [Mean (Standard Deviation); unit: mmHg/sec] — Rise of left ventricular pressure over time (dP/dT) produced by Multipoint pacing (MPP) in the peri-infarct region
  mmHg/sec | 1030.5 (92.63)
dP/dt produced by MPP in the remote myocardium [Mean (Standard Deviation); unit: mmHg/sec] — Rise of left ventricular pressure over time (dP/dT) produced by Multipoint pacing (MPP) in the remote myocardium
  mmHg/sec | 920.41 (44.42)
dP/dt produced by RV pacing [Mean (Standard Deviation); unit: mmHg/sec] — Rise of left ventricular pressure over time (dP/dT) produced by right ventricular pacing
  mmHg/sec | 893.03 (83.82)
dP/dt produced by CRT pacing in the peri-infarct region [Mean (Standard Deviation); unit: mmHg/sec] — Rise of left ventricular pressure over time (dP/dT) produced by CRT pacing in the peri-infarct region
  mmHg/sec | 945 (82.02)
dP/dt produced by CRT pacing in the remote myocardium [Mean (Standard Deviation); unit: mmHg/sec] — Rise of left ventricular pressure over time (dP/dT) produced by CRT pacing in the remote myocardium
  mmHg/sec | 1050.5 (7.78)

OUTCOME MEASURES:

1. Primary Outcome: Comparison of Acute Haemodynamic Response Produced by MPP in Peri-infarct Region and in the Remote Myocardium
Description: Comparison between
  1. percentage change of maximal left ventricular pressure over time (LV-dP/dTmax) produced by multipoint pacing (MPP) over spontaneous ventricular activation in the peri-infarct region and
  2. percentage change of maximal left ventricular pressure over time (LV-dP/dTmax) produced by multipoint pacing (MPP) over spontaneous ventricular activation in the remote myocardium
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: percentage change of dP/dT (mmHg/sec)
Arm/Group | Patients With Myocardial Scar
Number analyzed (Participants) | 2
percentage change of dP/dT (mmHg/sec) | 12.97 (0.95)

2. Primary Outcome: Comparison Between MPP and Standard CRT Pacing in Terms of Acute Haemodynamic Response
Description: Percentage change of LV dP/dT max produced by MPP over conventional single-site LV pacing in the peri-infarct region compared to the remote myocardium
  Comparison between
  1. percentage change of maximal left ventricular pressure over time (LV-dP/dTmax) produced by multipoint pacing (MPP) over conventional CRT pacing in the peri-infarct region and
  2. percentage change of maximal left ventricular pressure over time (LV-dP/dTmax) produced by multipoint pacing (MPP) over conventional CRT in the remote myocardium
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: percentage change of dP/dT (mmHg/sec)
Arm/Group | Patients With Myocardial Scar
Number analyzed (Participants) | 2
percentage change of dP/dT (mmHg/sec) | 13.49 (4.81)

ADVERSE EVENTS:
Time Frame: 1 day after the procedure
Arm/Group | Patients With Myocardial Scar
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-06): https://cdn.clinicaltrials.gov/large-docs/38/NCT04066738/Prot_SAP_000.pdf